CLINICAL TRIAL: NCT00099385
Title: Comprehensive Elementary School Risk Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Schonfeld, Director, Division of Developmental and Behavioral Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD045362 (NIH)
Record Dates: First submitted 2004-12-13; First posted 2004-12-14 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Risk Behavior
Keywords: social development; risk behaviors; social emotional education; classroom instruction
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Social Development Instruction — Weekly instruction during regular classroom time by classroom teacher using PATHS (Greenberg & Kusche) curriculum.

SUMMARY:
This project will evaluate the benefit of an enhanced social development program in grades 3-6 to decrease the onset of risky behaviors in pre-adolescents.

DETAILED DESCRIPTION:
Educational programs to promote the adoption of healthy behaviors and to decrease the onset of risky behaviors in pre-adolescents are far more likely to be successful than attempts to alter established patterns of high-risk behaviors. The project involves an evaluation of a comprehensive 4-year elementary school prevention initiative starting in 3rd grade. The prevention initiative, grounded in social cognitive, influence, and development theories is embedded within a pre-existing comprehensive elementary school social development program and will employ an evidence-based social skills curriculum (PATHS) in selected schools. The aim of the program is to teach children to use problem-solving and communication skills to negotiate and prevent high-risk behaviors.

Students attending schools that will receive the enhanced social development program will be compared to students attending schools that will receive the current, standard social development curriculum. The study hypothesizes that students who participate in the 4-year enhanced social development program will self-report fewer risk behaviors when surveyed by the school system in grades 6-8.

ELIGIBILITY:
Inclusion Criteria:

* All regular education students, including students in bilingual classes

Exclusion Criteria:

- Children attending special education classrooms.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2620 (Actual)
Dates: Start 2004-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Self reports of risky behaviors | Spring of 2008,2009,2010

SECONDARY OUTCOMES:
Academic test scores | annually 2006-2008
Measure of social problem solving skills: Social Problem Solving Dilemma | Spring 2007,2008

CONTACTS AND LOCATIONS:
Overall Officials: David J Schonfeld, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States